CLINICAL TRIAL: NCT02020941
Title: A Phase 2 Study of Carfilzomib and Bone Metabolism in Patients With Multiple Myeloma in First Relapse or Refractory to First Line Therapy
Brief Title: Carfilzomib in Treating Patients With Multiple Myeloma in First Relapse or Refractory to First-Line Therapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Attaya Suvannasankha (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Attaya Suvannasankha, Principal Investigator, Indiana University School of Medicine
Organization: Indiana University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IUCRO-0414; NCI-2013-01771 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); IUCRO-0414 (Other: Indiana University Cancer Center); P30CA082709 (NIH)
Record Dates: First submitted 2013-12-19; First posted 2013-12-25 (Estimated); Results first posted 2016-11-02 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-07

CONDITIONS: Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — carfilzomib; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (carfilzomib, dexamethasone) (Experimental): TREATMENT PHASE (COURSES 1-8): Patients receive carfilzomib IV over 30 minutes on days 1, 2, 8, 9, 15, and 16. Treatment repeats every 28 days for 8 courses in the absence of disease progression or unacceptable toxicity. Patients achieving less than PR also receive dexamethasone PO or IV weekly in courses 4-8.
  MAINTENANCE PHASE (COURSES 9-14): Patients receive carfilzomib IV over 30 minutes on days 1, 2, 15, and 16. Patients who received dexamethasone in the Treatment Phase continue to receive dexamethasone PO or IV weekly. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: carfilzomib; Drug: dexamethasone; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: carfilzomib — Given IV
  Other Names: Kyprolis; PR-171
Drug: dexamethasone — Given IV or PO
  Other Names: Aeroseb-Dex; Decaderm; Decadron; DM; DXM
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial studies how well carfilzomib works in treating patients with multiple myeloma in first relapse or refractory to first-line therapy. Carfilzomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the overall response rate of carfilzomib after 8 cycles of treatment in patients with first-relapsed myeloma.

SECONDARY OBJECTIVES:

I. To assess the overall response rate to single agent carfilzomib after 4 cycles of treatment.

II. To assess progression-free survival (PFS). III. To assess time to progression (TTP). IV. To assess duration of response (DOR). V. To assess toxicities.

TERTIARY OBJECTIVES:

I. To examine the effect of carfilzomib alone or in combination with dexamethasone on the following biologic end points and their correlation with response: measurements of bone remodeling (sodium fluoride F 18 positron emission tomography [PET], serum markers of bone remodeling and the bone marrow osteoblastic and osteoclastic differentiation and function) with the measurement of disease response and proteasome activity in the bone marrow microenvironment.

II. To describe recapture of response after progression in the maintenance phase.

OUTLINE:

TREATMENT PHASE (COURSES 1-8): Patients receive carfilzomib intravenously (IV) over 30 minutes on days 1, 2, 8, 9, 15, and 16. Treatment repeats every 28 days for 8 courses in the absence of disease progression or unacceptable toxicity. Patients achieving less than partial response (PR) also receive dexamethasone orally (PO) or IV weekly in courses 4-8.

MAINTENANCE PHASE (COURSES 9-14): Patients receive carfilzomib IV over 30 minutes on days 1, 2, 15, and 16. Patients who received dexamethasone in the Treatment Phase continue to receive dexamethasone PO or IV weekly. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Multiple myeloma (MM) in first relapse or refractory to first line therapy; the previous line of therapy should include either an immunomodulatory agent or a proteasome inhibitor

  * Refractory disease is defined as =< 25% response or progression during therapy or within 60 days after completion
  * The number of prior lines of anti-myeloma therapy will be determined as follows:

    * Induction chemotherapy for peripheral-blood stem cell harvest followed by planned mobilization and subsequent high-dose chemotherapy with autologous stem cell transplant (ASCT) is considered one therapy regardless of the induction regimen
    * Planned maintenance therapy after stem cell transplantation or other induction therapy is not considered a separate line of therapy, as long as there is no evidence of progression in the time between the induction or transplantation and the initiation of maintenance therapy
    * Two ASCTs within 6 months of each other is considered as one line unless different agents were used in the high-dose therapy-conditioning regimens
    * If the same regimen is repeated after a 6-month interval, they are considered to be two separate therapeutic lines
    * If cyclophosphamide is used for reasons other than planned stem cell mobilization, its use is considered to be a separate line of therapy
    * Dose modification of steroid and altering choices of steroid (i.e. from dexamethasone to prednisone) due to side effects, is not considered a line of therapy, as long as there is no evidence of progression
    * If a regimen was stopped for more than 2 months, its re-initiation is counted as another line of therapy
* Presence of existing lytic bone lesions either by skeletal X-ray, computed tomography (CT) scan or magnetic resonance imaging (MRI) scan
* Measurable MM disease, defined as one of the following:

  * A monoclonal immunoglobulin (Ig) concentration on serum electrophoresis of >= 0.5 g/dL for an IgG myeloma, >= 0.1 g/dL for an IgD myeloma or >= 0.5 g/dL for an IgA myeloma
  * Measurable urinary light chain secretion by quantitative analysis of >= 200 mg/24 hours
  * Involved serum free light chain (FLC) level >= 10 mg/dL, provided the serum FLC ratio is abnormal
  * Patients with oligo- or non-secretory disease must have bone marrow involvement with at least 30% plasmacytosis on aspiration
* Life expectancy >= 3 months as determined by the treating physician
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0, 1 or 2
* Absolute neutrophil count (ANC) >= 1.0 × 10^9/L (without transfusion support and without hematological growth factor support within 2 weeks of cycle 1 day 1)
* Platelets >= 50 × 10^9/L; if the bone marrow contains >= 50% plasma cells, a platelet count of >= 30 × 10^9/L is allowed (without transfusion support and without hematological growth factor support within 2 weeks of cycle 1 day 1)
* Aspartate aminotransferase (AST)/serum glutamic oxaloacetic transaminase (SGOT) and/or alanine aminotransferase (ALT)/serum glutamic pyruvic transaminase (SGPT) =< 2.5 × the upper limit of normal (ULN)
* Bilirubin < 2.0 mg/dL
* Serum creatinine =< 3.0 mg/dL or a calculated creatinine clearance of at least 15 mL/min (using the Cockcroft and Gault method)
* Adequate cardiac function defined as left ventricular ejection fraction (LVEF) >= 40%

  * NOTE: 2-dimensional (2-D) transthoracic echocardiogram (ECHO) is the preferred method of evaluation
  * Multigated acquisition scan (MUGA) is acceptable if ECHO is not available
* Written informed consent in accordance with federal, local, and institutional guidelines
* Females of childbearing potential (FCBP) must agree to ongoing pregnancy testing and to practice contraception; females are considered of childbearing potential unless they are surgically sterile (they have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are naturally postmenopausal for at least 12 consecutive months
* Male subjects must agree to practice contraception

Exclusion Criteria:

* No primary amyloidosis
* No plasma cell leukemia (> 2.0 × 10^9/L circulating plasma cells by standard differential)
* No treatment with an investigational product or device within 21 days of cycle 1 day 1
* No history of allergic reaction/hypersensitivity to any of the study medications, their analogues or excipients in the various formulations
* No treatment with cytotoxic therapy or monoclonal antibodies within 21 days prior to cycle 1 day 1
* No treatment with a steroid intended to treat myeloma within 14 days prior to cycle 1 day 1
* No autologous or allogeneic stem cell transplant within 3 months prior to cycle 1 day 1
* No radiotherapy within 21 days prior to cycle 1 day 1; however, if the radiation portal covered =< 5% of the bone marrow reserve, the patient may be enrolled irrespective of the end date of radiotherapy
* No major surgery within 14 days and minor surgery within 7 days prior to cycle 1 day 1
* No pregnant or lactating females
* No acute active infection requiring treatment (systemic antibiotics, antivirals, or antifungals) within 14 days prior to cycle 1 day 1
* No known human immunodeficiency virus (HIV) infection
* No active hepatitis B or C infection
* No unstable angina or myocardial infarction within 4 months prior to cycle 1 day 1, New York Heart Association (NYHA) class III or IV heart failure, uncontrolled angina, history of severe coronary artery disease, severe uncontrolled ventricular arrhythmias, sick sinus syndrome, or electrocardiographic evidence of acute ischemia or grade 3 conduction system abnormalities unless subject has a pacemaker
* No uncontrolled hypertension or uncontrolled diabetes (as determined by the treating physician) within 14 days prior to cycle 1 day 1
* No nonhematologic malignancy within the past 3 years with the exception of a) adequately treated basal cell carcinoma, squamous cell skin cancer, or thyroid cancer; b) carcinoma in situ of the cervix or breast; c) prostate cancer of Gleason grade 6 or less with stable prostate-specific antigen levels; or d) cancer considered cured by surgical resection or unlikely to impact survival during the duration of the study, such as localized transitional cell carcinoma of the bladder or benign tumors of the adrenal or pancreas
* No significant neuropathy (grades 3-4, or grade 2 with pain) within 14 days prior to cycle 1 day 1
* No known history of allergy to Captisol (a cyclodextrin derivative used to solubilize carfilzomib)
* No contraindication to any of the required concomitant drugs or supportive treatments, including hypersensitivity to all anticoagulation and antiplatelet options, antiviral drugs, or intolerance to hydration due to preexisting pulmonary or cardiac impairment
* No subjects with pleural effusions requiring thoracentesis or ascites requiring paracentesis within 14 days prior to cycle 1 day 1
* Any other clinically significant medical disease or condition that, in the Investigator's opinion, may interfere with protocol adherence or a subject's ability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-09; Primary Completion 2016-01 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Attaya Suvannasankha, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Indiana University Cancer Center, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This protocol was based on enrolling 23 patients. Due to slow accrual, the study was closed with 10 patients enrolled.
Groups:
- Treatment (Carfilzomib, Dexamethasone): TREATMENT PHASE (COURSES 1-8): Patients receive carfilzomib IV over 30 minutes on days 1, 2, 8, 9, 15, and 16. Treatment repeats every 28 days for 8 courses in the absence of disease progression or unacceptable toxicity. Patients achieving less than PR also receive dexamethasone PO or IV weekly in courses 4-8.
  MAINTENANCE PHASE (COURSES 9-14): Patients receive carfilzomib IV over 30 minutes on days 1, 2, 15, and 16. Patients who received dexamethasone in the Treatment Phase continue to receive dexamethasone PO or IV weekly. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.
  carfilzomib: Given IV
  dexamethasone: Given IV or PO
  laboratory biomarker analysis: Correlative studies
Period: Overall Study
Arm/Group | Treatment (Carfilzomib, Dexamethasone)
Started | 10
Completed | 2
Not Completed | 8
Not completed — Adverse Event | 1
Not completed — Physician Decision | 2
Not completed — Withdrawal by Subject | 1
Not completed — Disease Progression | 4

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Carfilzomib, Dexamethasone)
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.1 (6.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) After 8 Courses of Treatment
Description: : Evaluate the overall response rate of patients receiving therapy. Patients are considered as having a response if their overall response is Partial Response or better. The percentage of patients achieving this and the exact 95% confidence interval will be calculated. Responses will be defined using the International Myeloma Working Group-Uniform Response Criteria (IMWG-URC).
Time Frame: At 32 weeks
Population: All patients receiving at least one dose of study drug and having at least one evaluable post-baseline visit
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Carfilzomib, Dexamethasone)
Number analyzed (Participants) | 9
percentage of participants | 77.8 [40.0 to 97.2]

2. Secondary Outcome: Overall Response Rate (ORR) After 4 Courses of Treatment
Description: Evaluate the overall response rate of patients receiving therapy. Patients are considered as having a response if their overall response is Partial Response or better. The percentage of patients achieving this and the exact 95% confidence interval will be calculated. Responses will be defined using the International Myeloma Working Group-Uniform Response Criteria (IMWG-URC).
Time Frame: At 16 weeks
Population: All patients receiving at least one dose of study drug and having at least one evaluable post-baseline visit
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Carfilzomib, Dexamethasone)
Number analyzed (Participants) | 9
percentage of participants | 77.8 [40.0 to 97.2]

3. Secondary Outcome: Progression-free Survival (PFS)
Description: Analysis will be performed using Kaplan-Meier estimates. Time from date on treatment to date of progression for patients who progressed or date of death for patients who died without progressing. The observations of patients remaining alive and progression free were censored at date of last disease evaluation.
Time Frame: Time from first dose to first observed disease progression or death, assessed up to 2 years
Population: All patients enrolled and received treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Carfilzomib, Dexamethasone)
Number analyzed (Participants) | 10
months | 11.5 [2.9 to 16.4]

4. Secondary Outcome: Time to Progression (TTP)
Description: Analysis will be performed using Kaplan-Meier estimates. Time from date on treatment to date of progression. The observations of patients who died or remained alive and progression free were censored at date of death or last disease evaluation, respectively.
Time Frame: Time from first dose to disease progression, assessed up to 2 years
Population: All patients enrolled and received treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Carfilzomib, Dexamethasone)
Number analyzed (Participants) | 10
months | 11.5 [2.9 to 16.4]

5. Secondary Outcome: Duration of Response (DOR)
Description: Analysis will be performed using Kaplan-Meier estimates. Time from date of first confirmed response of partial response or better to date of progression or death. Only patients who had a response of partial response or better will be included in this analysis.
Time Frame: Time from first evidence of PR or better to disease progression or death, assessed up to 2 years
Population: All patients who had a response of partial response or better
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Carfilzomib, Dexamethasone)
Number analyzed (Participants) | 7
months | 8.9 [0.1 to 12.0]

6. Secondary Outcome: Treatment Related Adverse Events Grade 3 or Higher
Description: Number of unique patients who had a treatment related (possible, probable or definite) adverse events that were graded 3 or greater.
Time Frame: Up to 30 days after completion of study treatment, up to 2 years
Population: All patients enrolled and received treatment.
Measure: Number; unit: participants
Arm/Group | Treatment (Carfilzomib, Dexamethasone)
Number analyzed (Participants) | 10
participants | 5

ADVERSE EVENTS:
Time Frame: up to 2 years
Arm/Group | Treatment (Carfilzomib, Dexamethasone)
Serious Adverse Events (participants affected / at risk) | 2/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Carfilzomib, Dexamethasone) (N=10)
Heart Failure (Cardiac disorders) | 1
Lung infection (Infections and infestations) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Carfilzomib, Dexamethasone) (N=10)
Anemia (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Heart failure (Cardiac disorders) | 1
Ear pain (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Conjunctivitis (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Bloating (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 1
Dental caries (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 4
Flatulence (Gastrointestinal disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 4
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 3
Chills (General disorders) | 1
Edema limbs (General disorders) | 4
Fatigue (General disorders) | 3
Fever (General disorders) | 4
Flu like symptoms (General disorders) | 4
Infusion related reaction (General disorders) | 3
Irritability (General disorders) | 1
Pain (General disorders) | 1
Bronchial infection (Infections and infestations) | 1
Gum infection (Infections and infestations) | 1
Upper respiratory infection (Infections and infestations) | 4
Fall (Injury, poisoning and procedural complications) | 1
Neutrophil count decreased (Investigations) | 1
Platelet count decreased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Glucose intolerance (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ataxia (Nervous system disorders) | 1
Cognitive disturbance (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 2
Headache (Nervous system disorders) | 2
Nervous system disorders - Other (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 2
Tremor (Nervous system disorders) | 1
Depression (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Pelvic pain (Reproductive system and breast disorders) | 1
Reproductive system and breast disorders - Other (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash acneiform (Skin and subcutaneous tissue disorders) | 3
Skin ulceration (Skin and subcutaneous tissue disorders) | 1
Surgical and medical procedures - Other (Surgical and medical procedures) | 1
Flushing (Vascular disorders) | 1
Hypotension (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes